CLINICAL TRIAL: NCT05051917
Title: ITAlian Coronary Artery Aneurysm and Ectasia Observational Study in Patients With Acute Coronary Syndrome: The ITACA Registry
Brief Title: The Italian Coronary Artery Aneurysm and Ectasia In Patients With Acute Coronary Syndrome
Acronym: ITACA
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Collaborators: Fondazione GISE Onlus (Other)
Responsible Party: Principal Investigator, Giovanni Esposito, Professor of Cardiology, Federico II University
Other Study IDs: 22/21
Record Dates: First submitted 2021-09-15; First posted 2021-09-21 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Acute Coronary Syndrome; Angiographic Evidence if Coronary Aneurysms; Ectasia
Keywords: Aute Coronary Syndrome; Coronary Artery Artery; Ectasia
MeSH Terms: conditions — Acute Coronary Syndrome; Dilatation, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ITACA study is a prospective, observational no profit registry enrolling patients with Acute Coronary Syndrome and angiographic evidence of coronary aneurysms and/or ectasia.

DETAILED DESCRIPTION:
The ITACA study is aimed at evaluating short and long term outcomes in patients with acute coronary sindrome and angiographic evidence of coronary aneurysm and/or actasia. Data regarding safety and effectiveness of invasive and pharmacological treatment strategies will be also collected.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent;
* Patients aged ≥18 years;
* diagnosis of ACS (ST-elevation myocardial infarction, non ST-elevation myocardial infarction, unstable angina), in accordance with the definition provided in the latest guidelines;
* diagnosis of ectasia or coronary aneurysm according to the definitions contained in this protocol, either in the culprit vessel of the SCA than in another vessel. Coronary pseudoaneurysms are excluded.

Exclusion Criteria:

* impossibility or unwillingness to provide signed informed consent;
* contraindications to dual antiplatelet therapy;
* contraindications to anticoagulant therapy;
* active bleeding or severe anemia (Hb <6 g / dl);
* life expectancy <12 months;
* female patients with potential pregnancy;

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients undergoing coronary angiography with diagnosis of ACS and contextual detection of coronary ectasia or aneurysm in accordance with the definitions specified below. Patients with coronary pseudoaneurysms are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | two years
  A composite endpoint of myocardial infarction, stroke, cardiovascular death, myocardial revascularization and hospitalisation due to cardiovascular events

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Giuseppe Tarantino, Forlì, FC
  - Professor Giovanni Esposito, Naples

IPD SHARING:
Plan to Share IPD: No